CLINICAL TRIAL: NCT01042288
Title: A Phase II Trial of Carboplatin, Pemetrexed, and Panitumumab in Patients With Advanced Non-Squamous K-ras Wild Type Non-Small-Cell Lung Cancer
Brief Title: Carboplatin, Pemetrexed, and Panitumumab in Patients With Advanced Non-Squamous K-ras Wild Type NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 183
Record Dates: First submitted 2009-12-31; First posted 2010-01-05 (Estimated); Results first posted 2016-04-15 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-04

CONDITIONS: Non-Small-Cell Lung Cancer
Keywords: Non-Small-Cell Lung Cancer; NSCLC; Panitumumab; Vectibix; Pemetrexed; Alimta; Carboplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin; Pemetrexed; Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Carboplatin/Pemetrexed/Panitumumab (Experimental): Systemic Therapy
  Interventions: Drug: Carboplatin; Drug: Pemetrexed; Drug: Panitumumab

INTERVENTIONS:
Drug: Carboplatin — Carboplatin AUC=6IV, Day 1 of Cycles 1-6 (Cycles are 3 weeks / 21 days in length)
Drug: Pemetrexed — Pemetrexed 500mg/m² IV, Day 1 of Cycles 1-6 (Cycles are 3 weeks / 21 days in length)
  Other Names: Alimta
Drug: Panitumumab — Panitumumab 9mg/kg IV, Day 1 of Cycles 1-6 (Cycles are 3 weeks / 21 days in length)
  Other Names: Vectibix

SUMMARY:
The purpose of this multicenter, Phase II trial is to examine the role of a well-tolerated novel agent, panitumumab, in combination with a modern platinum doublet regimen using carboplatin and pemetrexed, in patients with advanced non-squamous wild type K-ras non-small-cell lung cancer (NSCLC). If this treatment proves to be well tolerated and associated with efficacy, this would provide rationale for further randomized studies.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years.
2. Histologically confirmed non-squamous NSCLC (squamous cell histology is ineligible). Cytologic specimens obtained by brushings, washings or needle aspiration of the defined lesion are acceptable. Sputum cytology alone is not acceptable. Mixed tumors with small cell elements are not eligible.
3. Newly diagnosed unresectable stage IIIB or stage IV disease. Patients with stage IIIB disease should be ineligible for combined modality therapy (i.e., pleural effusions, pericardial effusions, etc.).
4. At least one unidimensionally measurable lesion definable by magnetic resonance imaging (MRI) or computed tomography (CT) scan. Measurable disease is defined by the Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
5. Demonstration of K-ras wild type in archived tumor tissue. Tissue must be available for testing or results from previous K-ras testing must be available at the time of registration.
6. No prior antineoplastic chemotherapy for metastatic lung cancer. Patients may have received adjuvant treatment for stage I, II or III disease.
7. For patients who have had previous radiotherapy as definitive therapy for locally advanced NSCLC, recurrence must be outside of the original radiation therapy port. Radiation therapy must have been completed more than four weeks prior to study entry. Previous radiation must have covered < 30% of marrow bearing area.
8. Full recovery from surgery for patients who have undergone thoracotomy. Patients cannot start protocol treatment until at least three weeks after an operative procedure.
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
10. Life expectancy ≥ 12 weeks.
11. Normal bone marrow function within 7 days prior to initial treatment as defined by:

    * absolute neutrophil count (ANC) ≥1500/µL
    * platelets ≥100,000/µL
    * hemoglobin ≥8.0 g/dL. Patients may receive transfusions or erythropoietin to maintain or exceed this level.
12. Normal hepatic function as defined by:

    * bilirubin ≤1.5 x institutional upper limit of normal (ULN).
    * transaminases ≤2.5 x institutional ULN. In the presence of known hepatic metastases, transaminases may be ≤5 x institutional ULN.
13. Normal renal function within 7 days prior to initial treatment as defined by:

    * serum creatinine <2.0 mg/dL
    * estimated creatinine clearance (CrCl) ≥ 45 mL/min calculated by the Cockcroft-Gault method.
14. Normal metabolic function as follows:

    • Magnesium ≥ institutional lower limit of normal (LLN)
15. The ability to take folic acid, vitamin B12, and dexamethasone according to the protocol.
16. The ability to interrupt non-steroidal anti-inflammatory drugs (NSAIDs) 2 days before (5 days for long-acting NSAIDs), the day of, and 2 days following administration of pemetrexed.
17. Negative serum or urine pregnancy test within 7 days prior to initial study treatment.
18. Agreement of women of child-bearing potential (WOCBP) and men to use adequate contraception (hormonal or barrier method of birth control; abstinence) to prevent contraception during treatment and for a minimum of 6 months after the last study treatment.
19. Willingness and ability to comply with study and follow-up procedures.
20. Ability to understand the nature of this study and give written informed consent.

Exclusion Criteria:

1. NSCLC with squamous cell histology.
2. History of any invasive cancer treated within the previous 5 years with the exception of the disease under study, curatively treated non melanoma skin cancer or carcinoma in situ of the cervix.
3. Prior therapy which specifically and directly targets the EGFR pathway (e.g., cetuximab, gefitinib, erlotinib, lapatinib).
4. Active brain or meningeal metastases. Patients must have completed any previous radiotherapy at least four weeks prior to study entry and recovered from any toxicity associated with radiotherapy. Patients must have no on-going requirement for and must have discontinued corticosteroids.
5. Pregnancy or breast-feeding.
6. A serious active infection at the time of treatment or other serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
7. Acute hepatitis or known human immunodeficiency virus (HIV) infection.
8. Presence of third space fluid which is clinically significant and cannot be controlled by drainage.
9. History of interstitial lung disease (e.g., pneumonitis or pulmonary fibrosis or any evidence of interstitial lung disease on baseline chest CT scan).
10. History of any medical or psychiatric condition or laboratory abnormality that in the opinion of the investigator may increase the risks associated with the study participation or investigational product(s) administration or may interfere with the interpretation of the results.
11. Prior severe infusion reaction to a monoclonal antibody or history of allergic reactions attributed to compounds of similar chemical or biologic composition to agents used in study (e.g., carboplatin, pemetrexed).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-06; Primary Completion 2014-12 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David R Spigel, MD, Study Chair — SCRI Development Innovations, LLC
Locations (13):
- United States (13):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Hospital Cancer Institute, Orlando, Florida
  - Medical Oncology Associates of Augusta, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Baptist Hospital East, Louisville, Kentucky
  - Norton Cancer Institute, Louisville, Kentucky
  - Center for Cancer and Blood Disorders, Bethesda, Maryland
  - National Capital Clinical Research Consortium, Bethesda, Maryland
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Oncology Hematology Care, Cincinnati, Ohio
  - Cancer Centers of Southwest Oklahoma, Lawton, Oklahoma
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Peninsula Cancer Institute, Newport News, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One patient signed the consent but had a stroke prior to the pre-treatment and Cycle 1-Day 1 visits.
Period: Overall Study
Arm/Group | Carboplatin/Pemetrexed/Panitumumab
Started | 69
Maintenance | 27
Completed | 0 (Patients remained on maintenance until disease progression, toxicity or other reason to come off)
Not Completed | 69

BASELINE CHARACTERISTICS:
Arm/Group | Carboplatin/Pemetrexed/Panitumumab
Number analyzed (Participants) | 69
Age, Continuous [Median (Full Range); unit: years] | 65 [50 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 29
Region of Enrollment [Number; unit: participants]
  United States | 69

OUTCOME MEASURES:

1. Primary Outcome: Median Time to Progression (TTP)
Description: Defined as the time between Day 1-Cycle 1 and date of first documented disease progression assessed using Response Evaluation Criteria in Solid Tumors (RECISTS) v1.1.
Time Frame: 18 months
Population: All enrolled and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Pemetrexed/Panitumumab
Number analyzed (Participants) | 69
months | 6.11 [5.42 to 9.07]

2. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Defined as the time between Day 1-Cycle 1 and date of first documented disease progression or death.
Time Frame: Assessments by clinical evaluation, radiographic status, and date of disease progression, estimated 18 months
Population: All enrolled and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Pemetrexed/Panitumumab
Number analyzed (Participants) | 69
months | 5.75 [4.99 to 8.05]

3. Secondary Outcome: Median Overall Survival (OS)
Description: Defined as the time between Day 1-Cycle 1 to the date of death from any cause.
Time Frame: 18 months
Population: All enrolled and treated patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Carboplatin/Pemetrexed/Panitumumab
Number analyzed (Participants) | 69
months | 17.02 [11.33 to 19.68]

4. Secondary Outcome: Objective Response Rate
Time Frame: Projected 18 months
Population: All patients evaluated for response
Measure: Number; unit: percentage of evaluated participants
Arm/Group | Carboplatin/Pemetrexed/Panitumumab
Number analyzed (Participants) | 60
percentage of evaluated participants | 53

5. Secondary Outcome: Frequency of Adverse Events and Severity as a Measure of Toxicity
Description: Assessed using NCI CTCAE v4.0
Time Frame: Every 3 weeks (1 cycle) for 6 cycles, then every 7 weeks thereafter
Measure: Number; unit: participants
Arm/Group | Carboplatin/Pemetrexed/Panitumumab
Number analyzed (Participants) | 69
participants
  Rash | 55
  Nausea | 39
  Fatigue | 33
  Hypomagnesemia | 30
  Neutrophil Count Decreased | 30
  Platelet Count Decreased | 29
  Anemia | 28
  Mucositis | 23
  Dry Skin | 22
  Anorexia | 19
  Diarrhea | 19
  Constipation | 17
  White Blood Cell Decreased | 16
  Pruritus | 15
  Vomiting | 15
  Dehydration | 13
  Dysgeusia | 12
  Alopecia | 11

ADVERSE EVENTS:
Arm/Group | Carboplatin/Pemetrexed/Panitumumab
Serious Adverse Events (participants affected / at risk) | 24/69
Other Adverse Events (participants affected / at risk) | 67/69
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin/Pemetrexed/Panitumumab (N=69)
Abdominal pain (Gastrointestinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bladder infection (Infections and infestations) | 1
Cardiac disorders - Other, bradycardia (Cardiac disorders) | 1
Confusion (Psychiatric disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Duodenal Ulcer (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Fatigue (General disorders) | 1
Gastrointestinal disorders - Other, small bowel obstruction (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Infections and infestations - Other, bacteremia (Infections and infestations) | 1
Infections and infestations - Other, clostridium difficile infection (Infections and infestations) | 1
Infections and infestations - Other, Staphylococcus (Infections and infestations) | 1
Investigations - Other, pancytopenia (Investigations) | 1
Mucositis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Neutrophil count decreased (Investigations) | 1
Non-cardiac chest pain (General disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, COPD exacerbation (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1
Seizure (Nervous system disorders) | 2
stroke (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Thromboembolic event (Vascular disorders) | 2
Urinary Tract Infection (Infections and infestations) | 2
Urinary tract pain (Renal and urinary disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
White blood cell decreased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Carboplatin/Pemetrexed/Panitumumab (N=69)
rash (Skin and subcutaneous tissue disorders) | 55
Nausea (Gastrointestinal disorders) | 46
Fatigue (General disorders) | 43
Hypomagnesemia (Metabolism and nutrition disorders) | 36
platelet count decreased (Investigations) | 35
Anemia (Blood and lymphatic system disorders) | 33
neutrophil count decreased (Investigations) | 33
Constipation (Gastrointestinal disorders) | 28
diarrhea (Gastrointestinal disorders) | 25
Mucositis (Gastrointestinal disorders) | 25
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 24
Dry Skin (Skin and subcutaneous tissue disorders) | 22
Anorexia (Metabolism and nutrition disorders) | 20
Hyperglycemia (Metabolism and nutrition disorders) | 20
white blood cell decreased (Investigations) | 20
Pruritus (Skin and subcutaneous tissue disorders) | 19
Vomiting (Gastrointestinal disorders) | 19
Dehydration (Metabolism and nutrition disorders) | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 15
Hypokalemia (Metabolism and nutrition disorders) | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 14
Weight Loss (Investigations) | 14
Alopecia (Skin and subcutaneous tissue disorders) | 13
Dysgeusia (Nervous system disorders) | 12
abdominal pain (Gastrointestinal disorders) | 11
Edema limbs (General disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 9
rash acneiform (Skin and subcutaneous tissue disorders) | 9
alkaline phosphatase increased (Investigations) | 8
dizziness (Nervous system disorders) | 8
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 8
headache (Nervous system disorders) | 8
Hyponatremia (Metabolism and nutrition disorders) | 8
Insomnia (Psychiatric disorders) | 8
Fever (General disorders) | 7
Hyperkalemia (Metabolism and nutrition disorders) | 7
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7
Pain (General disorders) | 7
Alanine aminotransferase increased (Investigations) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 6
Chills (General disorders) | 6
creatinine increased (Investigations) | 6
dyspepsia (Gastrointestinal disorders) | 6
Investigations - Other, blood chloride decreased (Investigations) | 6
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 6
Skin and subcutaneous tissue disorders - Other, erythema (Skin and subcutaneous tissue disorders) | 6
Anxiety (Psychiatric disorders) | 5
Dry eye (Eye disorders) | 5
epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5
Infusion Related Reaction (General disorders) | 5
Investigations - Other, blood urea nitrogen decreased (Investigations) | 5
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5
Urinary Tract Infection (Infections and infestations) | 5
watering eyes (Eye disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4
Aspartate aminotransferase increased (Investigations) | 4
Blurred vision (Eye disorders) | 4
Bruising (Injury, poisoning and procedural complications) | 4
Eye pain (Eye disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 4
Hypotension (Vascular disorders) | 4
Investigations - Other, blood protein decreased (Investigations) | 4
Investigations - Other, creatinine decreased (Investigations) | 4
Investigations - Other, LDH increased (Investigations) | 4
Non-cardiac chest pain (General disorders) | 4
peripheral sensory neuropathy (Nervous system disorders) | 4
sinusitis (Infections and infestations) | 4
Skin infection (Infections and infestations) | 4
Thromboembolic event (Vascular disorders) | 4
Vaginal infection (Infections and infestations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites